CLINICAL TRIAL: NCT05660382
Title: Randomized, Double-blind, Phase III Study of the Efficacy and Safety of Miconazole Oil, Active Versus Placebo in the Treatment of Otomycosis
Brief Title: Phase III Efficacy and Safety Study of Miconazole Oil for Otomycosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hill Dermaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MZ-1015-ESP3-054
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis | interventions — Miconazole; Oils; Mineral Oil

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for participants, care providers, Investigators, outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Miconazole (2%) oil, administered as 5 drops per ear at ~30 mg per drop instilled into the external ear canal of the ear(s) affected by otomycosis, twice daily for 14 days.
  Interventions: Drug: Miconazole (2%) oil and mineral oil
- Placebo group (Placebo Comparator): Mineral oil, administered as 5 drops per ear instilled into the external ear canal of the ear(s) affected by otomycosis, twice daily for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Miconazole (2%) oil and mineral oil — Twice daily application, for 14 days.
  Other Names: Miconazole oil
  Arms: Active group
Other: Placebo — Twice daily application, for 14 days
  Other Names: Mineral oil
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to prove the that miconazole oil works well on fungal infections of the ears, by comparing the drug with a placebo. The researcher or the participants will not know if they are getting the drug or the placebo. The researcher will show the participants how to use the drug or placebo. After 14 days of using the drug or placebo, the participants will be examined by the researcher and graded on how well the drug worked on the ear(s) fungal infection. Participants will also be checked and asked for any bad side effects from the drug or the placebo.

DETAILED DESCRIPTION:
The purpose of this study is to gather confirmatory data on the efficacy and safety of 2% miconazole oil after topical otic administration in subjects with otomycosis, and to fully establish evidence of efficacy for miconazole oil compared to the placebo (mineral oil). A 14-day regimen of twice-daily administration of 2% miconazole oil will be compared with the same treatment regimen using the placebo, mineral oil. This study is a randomized, double-blind, parallel-group study to be conducted at up to 8 study centers in the US. An estimated 90 male or female subjects with otomycosis will receive study drug. Subjects will be randomly assigned in a 1:1 ratio within study site to receive miconazole oil or mineral oil for 14 days [administered as 5 drops per ear at ~30 mg per drop instilled into the external ear canal of the ear(s) affected by otomycosis]. Both the subject and the investigator and study staff will be blinded as to the contents of the study drug.

The primary efficacy endpoint is:

• Clinical Cure, defined as score of 0 for fungal elements, and for each of the signs/symptoms of pruritus, aural fullness and debris, at the Test of Cure visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females
2. Diagnosis of uncomplicated otomycosis of the external ear only, in the ear(s) that will be treated with study drug, with a score for fungal elements of 1 in each ear to be treated with study drug (see Section 7.4 for definitions of the scores for each of the otomycosis signs and symptoms). Subjects must also have the following signs and symptoms of otomycosis in the study ear: pruritus ≥2; debris ≥2; and aural fullness ≥2.
3. General good health as determined by medical examination and medical history, and who are free of clinically significant disease, including diabetes mellitus that is not well-controlled or that could interfere with the study
4. Females of childbearing potential must have had a negative urine pregnancy test at Screening/Baseline and must agree to use an effective method of contraception (as defined in Section 8.5) from Screening/Baseline up through the End of Treatment visit (see Section 6). Females of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >12 consecutive months). Females who are using oral, implanted, or injectable contraceptive hormones, an intrauterine device (IUD), barrier methods (diaphragm, condoms, spermicide) to prevent pregnancy, practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of childbearing potential
5. Subjects and/or their caregivers (as appropriate for the age of the subject) must have full legal capacity to volunteer
6. Subjects and/or their caregivers must have completed an appropriately administered institutional review board (IRB)-approved informed consent and assent (as applicable) prior to any study related procedures
7. Subjects and their caregivers (as applicable) must agree to comply with all requirements of the protocol
8. For subjects with only one ear meeting all study eligibility criteria, the subject will be eligible for the study, and the ear meeting all eligibility criteria will be treated with study drug and considered to be the study ear for the purposes of study evaluations. In case of bilateral otomycosis in which at least one ear meet all study eligibility criteria, the subject will be eligible for the study, both ears may be treated with study drug provided that both ears have a score of 1 for fungal elements, and the worse ear will be considered to be the study ear for the purposes of study evaluations. If both ears meet study eligibility criteria and are determined by the investigator to have the same degree of infection at Screening/Baseline, the left ear will be considered to be the study ear for the purposes of study evaluations.

Exclusion Criteria:

1. Any other dermatoses or conditions of the ear that may interfere with the evaluation of otomycosis, including concomitant otic infections (including bacterial infection) that require antimicrobial treatment, disease that has spread beyond the external ear(s), or pre-existing skin atrophy of the affected ear(s) that will be treated with study drug
2. Tympanostomy tube or perforated tympanic membrane in the ear(s) that will be treated with study drug
3. History of prior surgery directly affecting and compromising the external auditory canal and/or tympanic membrane of the ear(s) that will be treated with study drug, except for prior tympanostomy tube(s) that have already been removed and completely healed
4. Use of any topical medicated treatments for otomycosis within 14 days of study entry for the ear(s) that will be treated with study drug
5. Use of any systemic antifungal therapy within 28 days of study entry, warfarin within 28 days of study entry, immunosuppressive or immune-stimulating drugs within 28 days of study entry, or systemic steroids within 3 months of study entry
6. Fever of ≥100°F at study entry
7. Recurrent otomycosis that has been unresponsive to previous antifungal treatment within the last 12 months
8. Known hypersensitivity to any of the components in the test formulation
9. Participation in another investigative trial within 28 days of study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
primary efficacy endpoint | Day 22, test of cure
  Clinical Cure, defined as score of zero (0) for fungal elements and each of the signs/symptoms of pruritus, aural fullness and debris, at the Test of Cure visit.

SECONDARY OUTCOMES:
Clinical Cure at the End of Treatment | Day 15, end of treatment
  Score of zero (0) for fungal elements and for each signs/symptoms of otomycosis (debris, pruritus and aural fullness)
Modified Clinical Cure at Test of Cure | Day 22, test of cure
  Score of zero (0) for fungal elements, and score of "0" or "1" for each signs/symptoms of otomycosis (debris, pruritus and aural fullness)
Modified Clinical Cure at End of Treatment | Day 15, end of treatment
  Score of zero (0) for fungal elements, and score of "0" or "1" for each signs/symptoms of otomycosis (debris, pruritus and aural fullness)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Head and Neck Surgery Specialist, Chula Vista, California
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Charleston ENT Associates, LLC, North Charleston, South Carolina
  - Carolina ENT, Orangeburg, South Carolina
  - Spartanburg / Greer ENT & Allergy, Spartanburg, South Carolina
  - Alamo ENT Associates, San Antonio, Texas
  - ENT Center Of Utah, Salt Lake City, Utah